CLINICAL TRIAL: NCT01395121
Title: A Phase II Trial of Nilotinib in the Treatment of Patients With c-KIT Mutated Advanced Acral and Mucosal Melanoma
Brief Title: A Trial Looking at Nilotinib to Treat Acral and Mucosal Melanoma Skin Cancer That Has Spread
Acronym: NICAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2009/10020; 2009-012945-49 (EudraCT Number); Oxfordshire C 09/H0606/103 (Other: Main REC reference); CRUK/09/028 (Other: Cancer Research UK); CTA 15983/0226/001 (Other: MHRA); ISRCTN 39058880 (Other: ISRCTN)
Record Dates: First submitted 2011-04-13; First posted 2011-07-15 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Mucosal Lentiginous Melanoma; Acral Lentiginous Malignant Melanoma
Keywords: c-KIT mutation; advanced disease; tyrosine kinase inhibitors
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nilotinib (Experimental): nilotinib 400mgs oral tablets
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — nilotinib 400 mgs orally twice daily until disease progression or withdrawal from treatment
  Other Names: Tasigna

SUMMARY:
The aim of this study is to see if a drug called nilotinib (Tasigna®) is effective in the treatment of patients with a rare group of acral and mucosal melanomas that have a change (mutation) in a protein called cKIT. Nilotinib interferes with signalling inside cells with this mutation and it is believed that this may lead to shrinkage of tumours. Acral melanomas are found on the palms and soles and mucosal melanomas start inside body cavities rather than on the skin.

DETAILED DESCRIPTION:
NICAM has a two step consent process. Patients diagnosed with advanced acral or mucosal melanoma first consent for study registration and undergo screening tests including testing samples of melanoma tissue for the c-KIT mutation.

Following confirmation of the c-KIT mutation, patients are asked to consent to study entry with continuation of screening. Eligible patients then enter the study and commence taking nilotinib tablets twice a day for as long as clinical benefit is maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with c-KIT mutated histologically proven advanced mucosal or acral melanoma in which the mutation is not known to be associated with nilotinib resistance.
2. Advanced mucosal and acral melanoma defined as unresectable locally advanced or metastatic disease
3. The presence of one or more clinically or radiologically measurable lesions at least 10mm in size
4. Age 18 or greater
5. ECOG performance status 0, 1 or 2
6. Life expectancy greater than 12 weeks
7. At least 14 days since any major surgery
8. The capacity to understand the patient information sheet and ability to provide written informed consent
9. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
10. Women must not be pregnant or lactating with no intention of pregnancy during study treatment. Women of child bearing potential must have a negative serum pregnancy test prior to study entry (even if surgically sterilised). Men and women of childbearing potential must use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilisation) for the duration of the study and should continue such precautions for 6 months after receiving the last study treatment
11. Serum alanine transaminase (ALT) or serum aspartate aminotransferase ≤2.5 x upper limit of normal (ULN) and total serum bilirubin ≤1.5 x ULN
12. Serum creatinine ≤1.5 x ULN
13. Serum lipase and amylase <1.5 x ULN
14. Haemoglobin ≥9.0 g/dL, absolute neutrophil count ≥1.5 x 109/L, platelets ≥100 x 109/L
15. Prothrombin time (PT) ≤1.5 x ULN
16. Able to swallow and retain oral medication.

Exclusion Criteria:

1. Intracranial disease, unless there has been radiological evidence of stable intracranial disease > 6 months. In the case of a solitary brain metastasis, evidence of a disease-free interval of at least 3 months post surgery. All patients previously treated for brain metastases must be stable off corticosteroid therapy for at least 28 days
2. Women who are pregnant, nursing, or planning to become pregnant during the course of the trial
3. Men who plan to father a child during the course of the trial
4. Use of any investigational drug within 30 days prior to screening (both cancer and non cancer treatments)
5. Use of herbal or chinese medication
6. Use of therapeutic coumarin derivatives (ie warfarin, acenocoumarol, phenprocoumon)
7. Significant cardiac disease including patients who have or who are at significant risk of developing prolongation of QTc
8. Severe and/or uncontrolled medical disease
9. Known chronic liver disease
10. Past medical history of chronic pancreatitis
11. Known HIV infection
12. Previous radiotherapy to 25% or more of the bone marrow
13. Radiation therapy in the 4 weeks prior to study entry
14. Prior exposure to a tyrosine kinase inhibitor
15. Known lactose intolerance
16. Any malabsorption syndrome (i.e. partial gastrectomy, small bowel resection, Crohn's disease or ulcerative colitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with the c-KIT mutation who remain progression free at 6 months. | 6 months
  Progression free survival times will be measured from the date of enrolment into the treatment phase until the first date (following start of treatment) of either death or confirmed progressive disease according to RECIST.

SECONDARY OUTCOMES:
toxicity of treatment | evaluated every 4 weeks whilst the patient is on treatment (on average estimated to be between 4 and 52 weeks)
  Treatment related toxicity will be assessed at each clinic visit approximately every 4 weeks whilst the patient continues on study treatment. Study treatment will continue until the patient relapses or is withdrawn from study therapy (on average estimated to be between 4 and 52 weeks).
response at 12 weeks | tumours measured at 12 weeks from start of treatment
  Lesions must be measured and or evaluated at 12 weeks in accordance with the Response evaluation criteria in solid tumours (RECIST)
overall survival | Expected to be 6 - 12 months (Measured from commencement of treatment until time of death)

CONTACTS AND LOCATIONS:
Overall Officials: James Larkin, MA BM BCh MRCP PhD, Principal Investigator — Royal Marsden NHS Foundation
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom